CLINICAL TRIAL: NCT02393976
Title: NUTRITIONAL EFFECTS AND INFLUENCE IN THE MORBIDITY AND MORTALITY OF DIET IMMUNOMODULATORY IN FAST-TRACK SURGERY
Brief Title: IMMUNONUTRITION IN FAST-TRACK SURGERY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Collaborators: Fundación Mutua Madrileña (Other)
Responsible Party: Principal Investigator, Pedro Moya, PHD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: Cirugía2
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Last update posted 2015-03-20 (Estimated); Status verified 2015-03

CONDITIONS: IMMUNONUTRITION
MeSH Terms: interventions — Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CONTROL (Other): STANDARD NUTRITION
  Interventions: Dietary Supplement: STANDART NUTRITION
- IMMUNONUTRITION (Experimental): INMUNONUTRITION
  Interventions: Dietary Supplement: IMMUNONUTRITION

INTERVENTIONS:
Dietary Supplement: IMMUNONUTRITION — IMMUNONUTRITION SUPLEMENTS PERIOPERATIVE
  Arms: IMMUNONUTRITION
Dietary Supplement: STANDART NUTRITION — STANDART NUTRITION PERIOPERATIVE
  Arms: CONTROL

SUMMARY:
Compare the results in terms of morbidity, mortality and hospitalization among patients with input from immunonutrients and patients with enteral nutrition intake of high calorie and high protein undergoing colorectal surgery within a multimodal rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing colorectal surgery.
* Signing informed consent.

Exclusion Criteria:

* Patients with no oral nutrition (dysphagia, esophageal stricture, pyloric stenosis)
* Patients with contraindications for electrical stimulation.
* Psychiatric Disorders
* HIV
* Pregnant or breastfeeding
* intestinal obstruction
* uncontrolled infection
* ASA IV
* No acceptance or failure to follow protocol multimodal rehabilitation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Infectious complications | UP TO 30 DAYS POST-OPERATIVE

CONTACTS AND LOCATIONS:
Locations (1):
- Pedro Moya, Elche, Alicante, Spain

REFERENCES:
- [Derived] Moya P, Soriano-Irigaray L, Ramirez JM, Garcea A, Blasco O, Blanco FJ, Brugiotti C, Miranda E, Arroyo A. Perioperative Standard Oral Nutrition Supplements Versus Immunonutrition in Patients Undergoing Colorectal Resection in an Enhanced Recovery (ERAS) Protocol: A Multicenter Randomized Clinical Trial (SONVI Study). Medicine (Baltimore). 2016 May;95(21):e3704. doi: 10.1097/MD.0000000000003704. PMID 27227930